CLINICAL TRIAL: NCT02122458
Title: Blast-exposed Veterans With Auditory Complaints
Brief Title: Blast Exposed Veterans With Auditory Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1164-R
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hearing Impairment; Hearing Aid Fitting
Keywords: hearing impairment; post-traumatic stress disorder; traumatic brain injury; auditory processing disorder
MeSH Terms: conditions — Hearing Loss; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Auditory Perceptual Disorders | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: The primary study was diagnostic, with a goal of better understanding and determining the best diagnostic assessment battery for capturing the hearing and auditory problems reported by blast-exposed Veterans. The secondary purpose was to implement a preliminary treatment study to determine if blast-exposed Veterans with hearing complaints, but normal audiometric data benefited from low-gain hearing aids. This secondary treatment study is the clinical trial portion of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (7):
- Immediate Hearing Aid Treatment: Blast-exposed Only (Active Comparator): This group consisted of blast-exposed Veterans with auditory complaints but normal audiometric test results. These Veterans were negative for significant PTSD. They were fitted with open-fit hearing aids that provided mild high-frequency amplification and were monitored for 6 months.
  Interventions: Device: mild-gain hearing aids with high-frequency emphasis over 6-months
- Immediate Hearing Aid Treatment: Blast-exposed with PTSD (Active Comparator): This group consisted of blast-exposed Veterans with auditory complaints but normal audiometric test results. These Veterans were comorbid for significant PTSD. They were fitted with open-fit hearing aids that provided mild high-frequency amplification and were monitored for 6 months.
  Interventions: Device: mild-gain hearing aids with high-frequency emphasis over 6-months
- Delayed Hearing Aid Treatment: Blast-exposed Only (Active Comparator): This group consisted of blast-exposed Veterans with auditory complaints but normal audiometric test results. These Veterans were negative for significant PTSD. They were fitted with hearing aids after a 6-month delay. Their performance was monitored 6-months pre-fitting and for the 6 months after the fitting.
  Interventions: Device: mild-gain hearing aids with high-frequency emphasis over 6-months
- Non-treatment Diagnostic Testing: Normal (No Intervention): This group consisted of Veterans who completed the same pre-treatment diagnostic testing as the three treatment groups but were not enrolled in the hearing aid treatment protocol. This group included neurotypical Veterans with normal hearing and were negative for blast-exposure and PTSD.
- Non-Treatment Diagnostic Testing: Blast-exposed Only (No Intervention): This group consisted of Veterans who completed the same pre-treatment diagnostic testing as the three treatment groups but were not enrolled in the hearing aid treatment protocol. This group consisted of blast-exposed Veterans with auditory complaints but normal audiometric test results. They were negative for significant PTSD.
- Non-treatment Diagnostic Testing: Blast-exposed with PTSD (No Intervention): This group consisted of Veterans who completed the same pre-treatment diagnostic testing as the three treatment groups but were not enrolled in the hearing aid treatment protocol. This group consisted of blast-exposed Veterans with auditory complaints but normal audiometric test results. These Veterans were comorbid for significant PTSD.
- Non-treatment Diagnostic Testing: PTSD Only (No Intervention): This group consisted of Veterans who completed the same pre-treatment diagnostic testing as the three treatment groups but were not enrolled in the hearing aid treatment protocol. This group was negative for blast-exposure and hearing loss but positive for significant PTSD.

INTERVENTIONS:
Device: mild-gain hearing aids with high-frequency emphasis over 6-months — open-fit hearing aids with mild amplification in the high frequencies.
  Other Names: hearing aids
  Arms: Delayed Hearing Aid Treatment: Blast-exposed Only; Immediate Hearing Aid Treatment: Blast-exposed Only; Immediate Hearing Aid Treatment: Blast-exposed with PTSD

SUMMARY:
The purpose of this study is to study blast-exposed Veterans who report hearing handicap but show normal or near normal results on standard audiometric testing. The characteristics and nature of their auditory and auditory-related skills will be examined, along with whether coexisting PTSD contributes to the hearing problems of these Veterans. In a preliminary treatment study, a sub-sample of these Veterans will be fitted with mild-gain hearing aids to determine if they benefit from low-level amplification of high-frequency sounds.

DETAILED DESCRIPTION:
The purpose of this study is to study blast-exposed Veterans who report hearing handicap but show normal or near normal results on standard audiometric testing. The characteristics and nature of their auditory and auditory-related skills will be examined with a battery of behavioral and physiologic measures. The potential contributions of co-occurring PTSD also will be evaluated. In a preliminary treatment study, a sub-sample of the targeted Veterans will be fitted with mild-gain hearing aids to determine if they benefit from low-level amplification of high-frequency sounds.

This study consists of two parts. In Part 1, four groups of Veterans, aged 20 - 50 years, will complete a battery of auditory and auditory-related assessments to better understand the deficit sources and patterns. The assessment measures will consist of questionnaires, behavioral tests, and auditory physiologic measures. One group will consist of blast-exposed Veterans with auditory problems but no PTSD. The second group will consist of blast-exposed Veterans with auditory problems plus PTSD. The third group will consist of Veterans with PTSD but no reported auditory problems, and the fourth groups will be a normal control group.

In Part 2 of the study (clinical trial portion), a smaller group of participants from the first and second groups will be fitted with mild-gain open-fit hearing aids to determine if they benefit from mild high-frequency amplification. Changes in hearing handicap and speech perception will be compared from baseline to 6-months post-fitting. Perceived hearing aid benefit, hearing aid use time, and intent to continue use will be measured at the end of a 6-month treatment period. A delayed treatment group will be formed from group 1 and will be followed over a 12-month period with hearing aids fitted at 6 months. The participants will be assigned randomly from Part 1 of the study.

The information obtained from this study will help us understand the auditory problems experienced by blast-exposed Veterans and eventually contribute to the development of an efficient and effective assessment battery and intervention approaches.

ELIGIBILITY:
Inclusion Criteria:

* age 20 - 50 years; U.S. Veteran;
* English-speaking;
* history of blast exposure and no history of blast exposure;
* history of PTSD and no history of PTSD;
* self-perceived hearing handicap and no self-perceived hearing handicap;
* normal or near normal pure tone hearing thresholds;
* history of brain injury and no history of brain injury;
* normal vision.

Exclusion Criteria:

* hyperacusis;
* marked tinnitus;
* pure tone hearing thresholds consistent with a hearing loss;
* greater the 20/30 vision screening results (corrected or uncorrected);
* marked speech perception deficits

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 363 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila R Pratt, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (3):
- United States (3):
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Sioux Falls VA Health Care System, Sioux Falls, SD, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual participant data and the study data dictionary will be made available upon request to the PI (spratt@pitt.edu).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the conclusion of the study and after publication of planned study manuscripts. The time will not be limited.
Access Criteria: Those requesting data will need to provide a plan for how the data will be used.

REFERENCES:
- [Background] Gallun FJ, Papesh MA, Lewis MS. Hearing complaints among veterans following traumatic brain injury. Brain Inj. 2017;31(9):1183-1187. doi: 10.1080/02699052.2016.1274781. PMID 28981349
- [Background] Gallun FJ, Lewis MS, Folmer RL, Diedesch AC, Kubli LR, McDermott DJ, Walden TC, Fausti SA, Lew HL, Leek MR. Implications of blast exposure for central auditory function: a review. J Rehabil Res Dev. 2012;49(7):1059-74. doi: 10.1682/jrrd.2010.09.0166. PMID 23341279
- [Background] Koerner TK, A Papesh M, Gallun FJ. A Questionnaire Survey of Current Rehabilitation Practices for Adults With Normal Hearing Sensitivity Who Experience Auditory Difficulties. Am J Audiol. 2020 Dec 9;29(4):738-761. doi: 10.1044/2020_AJA-20-00027. Epub 2020 Sep 23. PMID 32966118
- [Background] Folmer RL, Billings CJ, Diedesch-Rouse AC, Gallun FJ, Lew HL. Electrophysiological assessments of cognition and sensory processing in TBI: applications for diagnosis, prognosis and rehabilitation. Int J Psychophysiol. 2011 Oct;82(1):4-15. doi: 10.1016/j.ijpsycho.2011.03.005. Epub 2011 Mar 16. PMID 21419179
- [Background] Papesh MA, Stefl AA, Gallun FJ, Billings CJ. Effects of Signal Type and Noise Background on Auditory Evoked Potential N1, P2, and P3 Measurements in Blast-Exposed Veterans. Ear Hear. 2021 Jan/Feb;42(1):106-121. doi: 10.1097/AUD.0000000000000906. PMID 32520849
- [Background] Hoover EC, Souza PE, Gallun FJ. Auditory and Cognitive Factors Associated with Speech-in-Noise Complaints following Mild Traumatic Brain Injury. J Am Acad Audiol. 2017 Apr;28(4):325-339. doi: 10.3766/jaaa.16051. PMID 28418327
- [Background] Gallun FJ, Diedesch AC, Kubli LR, Walden TC, Folmer RL, Lewis MS, McDermott DJ, Fausti SA, Leek MR. Performance on tests of central auditory processing by individuals exposed to high-intensity blasts. J Rehabil Res Dev. 2012;49(7):1005-25. doi: 10.1682/jrrd.2012.03.0038. PMID 23341276
- [Background] Fausti SA, Wilmington DJ, Gallun FJ, Myers PJ, Henry JA. Auditory and vestibular dysfunction associated with blast-related traumatic brain injury. J Rehabil Res Dev. 2009;46(6):797-810. doi: 10.1682/jrrd.2008.09.0118. PMID 20104403
- [Background] Reavis KM, Snowden JM, Henry JA, Gallun FJ, Lewis MS, Carlson KF. Blast Exposure and Self-Reported Hearing Difficulty in Service Members and Veterans Who Have Normal Pure-Tone Hearing Sensitivity: The Mediating Role of Posttraumatic Stress Disorder. J Speech Lang Hear Res. 2021 Nov 8;64(11):4458-4467. doi: 10.1044/2021_JSLHR-20-00687. Epub 2021 Sep 28. PMID 34582257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited through flyers, letters, VA audiologists, and Veteran organizations. Recruitment activities occurred Year 1 through Year 4 of the study.
  It should be noted that the participants enrolled in the hearing aid treatment arms (clinical trial portion of the study) completed diagnostic testing prior to completing the hearing aid treatment. The remaining participants only completed the diagnostic testing (Non-treatment Diagnostic Testing).
Pre-assignment Details: Preliminary testing and review of clinical records excluded 137 participants prior to group assignment.
Period: Overall Study
Arm/Group | Immediate Hearing Aid Treatment: Blast-exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only | Non-treatment Diagnostic Testing: Normal | Non-treatment Diagnostic Testing: Blast-exposed Only | Non-treatment Diagnostic Testing: Blast-exposed With PTSD | Non-treatment Diagnostic Testing: PTSD Only
Started | 12 | 18 | 7 | 82 | 45 | 43 | 19
Completed | 9 | 13 | 7 | 67 | 31 | 23 | 18
Not Completed | 3 | 5 | 0 | 15 | 14 | 20 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 4 | 4 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0 | 7 | 5 | 15 | 1
Not completed — Did not qualify at initial testing or after chart review | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Experimental Error | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Deployed or Moved | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Scheduling Delays - Unable to Complete | 0 | 1 | 0 | 4 | 1 | 1 | 0
Not completed — Noncompliance | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Veterans between the ages of 20 and 50 years of age who had normal hearing on standard audiometric testing, who had significant or no self-reported hearing handicap, significant or no history of blast-exposure, significant or no PTSD, normal vision and no history of prior brain injuries or diseases that were not blast-related. Preliminary testing and review of clinical records excluded 137 participants. These participants are not included in the baseline participant numbers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Hearing Aid Treatment: Blast-exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only | Non-treatment Diagnostic Testing: Normal | Non-treatment Diagnostic Testing: Blast-exposed Only | Non-treatment Diagnostic Testing: Blast-exposed With PTSD | Non-Treatment Diagnostic Testing: PTSD Only | Total
Number analyzed (Participants) | 12 | 18 | 7 | 82 | 45 | 43 | 19 | 226
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.01 (8.63) | 37.46 (6.73) | 39.21 (8.47) | 35.23 (8.29) | 35.32 (6.72) | 34.52 (6.42) | 34.85 (8.10) | 37.08 (7.77)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Participants by Sex: Number of Male Participants Per Arm | 10 | 15 | 7 | 56 | 39 | 38 | 10 | 175
  Participants by Sex: Number of Female Participants Per Arm | 2 | 3 | 0 | 26 | 6 | 5 | 9 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 8 | 5 | 4 | 1 | 21
  Not Hispanic or Latino | 10 | 17 | 7 | 73 | 40 | 39 | 18 | 204
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 4
  Asian | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 0 | 2 | 14 | 2 | 5 | 1 | 26
  White | 10 | 15 | 3 | 56 | 40 | 32 | 16 | 172
  More than one race | 0 | 1 | 0 | 9 | 3 | 4 | 1 | 18
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 18 | 7 | 82 | 45 | 43 | 19 | 226
Age [Mean (Full Range); unit: Years] | 37.01 [26.4 to 50.6] | 37.46 [27.7 to 49.1] | 39.21 [28.3 to 50.9] | 35.23 [20.6 to 50.9] | 35.32 [23.2 to 49.9] | 34.52 [23.4 to 48.6] | 34.85 [25.10 to 49.10] | 37.08 [20.6 to 50.9]

OUTCOME MEASURES:

1. Primary Outcome: Hearing Handicap Inventory for Adults (HHIA)
Description: Self-perceived hearing handicap was measured with the Hearing Handicap Inventory for Adults (HHIA), pre- and 6-months post-hearing aid fitting. The minimum score is 0 and the maximum score is 100, with the higher score reflecting greater handicap (worse outcome). The data are presented as a comparison between the two questionnaire administrations (pre- and 6-months post-fitting). The null hypothesis tested was that there would be no difference between the HHIA administered at baseline (pre-fitting) and 6-months post-fitting for all groups.
Time Frame: The participants wore their hearing aids for 6 months-fitting (baseline to 6-months post-fitting). The delayed group had a 6-month delay prior to treatment.
Population: A total of 37 participants were recruited to enroll in the treatment (clinical trial) part of the study. Eight of these 37 participants did not complete the treatment. The handicap scale was administered twice (pre-fitting and 6-months post-fitting) to the three groups. The Outcome Measure Data Table reflect comparisons between the overall scores for the 2 questionnaire administrations.
Measure: Mean (95% Confidence Interval); unit: Scale score
Arm/Group | Immediate Hearing Aid Treatment: Blast-exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only
Number analyzed (Participants) | 9 | 13 | 7
Scale score | 26.20 [19.04 to 33.33] | 37.34 [31.37 to 43.32] | 19.21 [10.48 to 27.95]
Statistical Analysis 1: Comparison: Immediate Hearing Aid Treatment: Blast-exposed Only vs Immediate Hearing Aid Treatment: Blast-exposed With PTSD vs Delayed Hearing Aid Treatment: Blast-exposed Only; The null hypothesis evaluated by the HHIA was that self-perceived hearing handicap would not reduce from baseline to 6-months post-fitting; Test type: Superiority; p = .05, Mixed Models Analysis — Given the preliminary nature of this treatment study and the small number of participants the p-value was not adjusted for multiple comparisons; An Adjusted Rank Transform was applied to the data prior to applying the mixed model analyses; Mean Difference (Net) = .448, 95% CI 2-sided [-8.66 to 9.56]

2. Primary Outcome: Hearing Aid Benefit (Abbreviated Profile of Hearing Aid Benefit, APHAB)
Description: The Abbreviated Profile of Hearing Aid Benefit (APHAB) was administered at the end of the treatment period (6-months post-fitting) to measure self-perceived benefit. The APHAB is a 24-item self-assessment inventory used to indicate the extent to which listeners experience listening difficulties (with and without hearing aids) in various settings. The questionnaire uses a 7-point scale that corresponds to the frequency with which difficulties are experienced (99 to 1% of the time). The APHAB was administered for both unaided listening and aided listening, and benefit was calculated by subtracting the mean aided scores from the mean unaided scores. Higher benefit scores (e.g., 99% unaided - 25% aided vs. 99% unaided - 50% aided) reflected greater benefit (better outcome) and negative scores were possible. The null hypothesis tested was that no hearing aid benefit would be demonstrated by any of the 3 groups at 6-months post-fitting.
Time Frame: The APHAB was administered 6-months post-fitting. The delayed group had a 6-month delay prior to the treatment (6-months of wearing the hearing aids).
Population: A total of 37 participants were recruited to enroll in the treatment (clinical trial) part of the study. Eight of these 36 participants did not complete the treatment. The APHAB benefit data shown here were collected at 6-months post-fitting (end of the treatment) from the 3 groups of participants. One APHAB (aided and unaided portions) was completed per participant.
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Immediate Hearing Aid Treatment: Blast-Exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only
Number analyzed (Participants) | 9 | 13 | 7
Scale score | -.362 (.301) | -.270 (.821) | -.080 (.331)
Statistical Analysis 1: Comparison: Immediate Hearing Aid Treatment: Blast-Exposed Only vs Immediate Hearing Aid Treatment: Blast-exposed With PTSD vs Delayed Hearing Aid Treatment: Blast-exposed Only; Test type: Superiority; p = .05, ANOVA — Given the small sample size and the preliminary nature of this study, the p-value was not adjusted for multiple comparisons

3. Primary Outcome: Intent to Continue Use
Description: The participants reported whether they would continue to use their hearing aids after the study has ended. The null hypothesis tested was that neither group would demonstrate a significant preference for retaining their hearing aids.
Time Frame: 6 months post-fitting
Population: A total of 37 participants were recruited to enroll in the treatment (clinical trial) part of the study. Eight of these 36 participants did not complete the treatment. The data shown here were collected at 6-months post-fitting (end of the treatment) from the 3 groups of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Hearing Aid Treatment: Blast-Exposed Only | Immediate Hearing Aid Treatment: Blast-Exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only
Number analyzed (Participants) | 9 | 13 | 7
Participants | 9 | 13 | 7

4. Secondary Outcome: Hearing Aid Use Time (Number of Participants With an Average Hearing Aid Use Time of 4 Hours a Day)
Description: Hearing aid use time was the number of participants who wore their hearing aids for an average of at least 4 hours per day. The average number of hours that the participants used their hearing aids was measured by their hearing aid data logging systems. These data were collected at the end of the treatment interval for each participant and were considered a positive outcome if they wore their hearing aids at least 4 hours a day on average after 1 month of use. The null hypothesis tested was that none of the participants in the three groups would not demonstrate hearing aid use time 4 hours or more, on average per day.
Time Frame: Hearing aid use time was collected at 6 months post-fitting.
Population: These data are a count of participants who wore their hearing aids at least 4 hours per day on average after 1 month of use. A total of 37 participants were recruited to enroll in the treatment (clinical trial) part of the study. Eight of these 37 participants did not complete the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Hearing Aid Treatment: Blast-exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only
Number analyzed (Participants) | 9 | 13 | 7
Participants | 9 | 7 | 3

5. Secondary Outcome: Speech Perception in Quiet and in Noise
Description: The participants' speech perception was measured at the word level with the California Consonant Test (CCT). The CCT is a 50 item a closed-set word identification test. It was administered at 3 timepoints (pre-fitting, 1-week post-fitting, and 6-months post-fitting), with testing was completed in quiet and in background noise (speech babble, +3 dB signal/babble) at each timepoint. The participants were unaided during the pre-fitting testing but wore their hearing aids during the two post-fitting sessions. The outcome measure was the proportion of correct trials out of 50. A correct trial consisted of an accurate identification of the target word presented to the participant in the sound-field at 40 dB sensation level. The null hypothesis tested was that speech perception would not improve over the treatment intervals for the groups for either test condition (quiet and noise).
Time Frame: The CCT was administered immediately pre-fitting (unaided), 1 week post-fitting (aided), and 6 months post-fitting (aided).
Population: A total of 37 participants were recruited to enroll in the treatment (clinical trial) part of the study. Eight of these 37 participants did not complete the treatment and are not reflected in the data reported here.
Measure: Mean (Standard Deviation); unit: Proportion Correct
Arm/Group | Immediate Hearing Aid Treatment: Blast-exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only
Number analyzed (Participants) | 9 | 13 | 7
Proportion Correct
  Pre-fitting Score in Quiet | .92 (.017) | .93 (.013) | .95 (.018)
  Pre-fitting Score in Noise | .69 (.044) | .73 (.033) | .72 (.047)
  1-week Post-fitting Test Score in Quiet | .96 (.018) | .93 (.014) | .95 (.019)
  1-week Post-fitting Test Score in Noise | .83 (.046) | .79 (.035) | .79 (.049)
  Final Test Score in Quiet | .96 (.009) | .95 (.007) | .95 (.010)
  Final Test Score in Noise | .84 (.037) | .82 (.028) | .71 (.040)

ADVERSE EVENTS:
Time Frame: Adverse events were queried for each individual participant per session from enrollment to completion of their participation in study and summarized yearly at IRB renewal, Adverse Events were collected for 6 months from all participants except for those enrolled in the Delayed Hearing Aid Treatment Arm/Group, which was assessed for up to 1 year.
Description: This was a minimal risk study, so adverse events were not expected but recorded and reported if they occurred or were reported by participants.
Arm/Group | Immediate Hearing Aid Treatment: Blast-exposed Only | Immediate Hearing Aid Treatment: Blast-exposed With PTSD | Delayed Hearing Aid Treatment: Blast-exposed Only | Non-treatment Diagnostic Testing: Normal | Non-treatment Diagnostic Testing: Blast-exposed Only | Non-treatment Diagnostic Testing: Blast-exposed With PTSD | Non-treatment Diagnostic Testing: PTSD Only
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/18 | 0/7 | 0/82 | 0/45 | 0/43 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/18 | 0/7 | 0/82 | 0/45 | 0/43 | 0/19
Other Adverse Events (participants affected / at risk) | 0/12 | 0/18 | 0/7 | 0/82 | 0/45 | 0/43 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Hearing Aid Treatment: Blast-exposed Only (N=12) | Immediate Hearing Aid Treatment: Blast-exposed With PTSD (N=18) | Delayed Hearing Aid Treatment: Blast-exposed Only (N=7) | Non-treatment Diagnostic Testing: Normal (N=82) | Non-treatment Diagnostic Testing: Blast-exposed Only (N=45) | Non-treatment Diagnostic Testing: Blast-exposed With PTSD (N=43) | Non-treatment Diagnostic Testing: PTSD Only (N=19)
Middle ear infection and mass (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One participant acquired an ear infection that required referral for medical intervention. The infection failed to resolve and eventually a middle ear mass was diagnosed. The participant was withdrawn

LIMITATIONS AND CAVEATS:
The hearing aid treatment portion of this study was preliminary in nature and limited by the number of participants enrolled and amount of time with which those enrolled wore their hearing aids. Problems with hearing aid wear-time compliance limited interpretation and applicability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT02122458/Prot_SAP_000.pdf